CLINICAL TRIAL: NCT03954548
Title: Prospective, Randomized, Multicenter, Tandem Study Evaluating the Safety and Effectiveness of the CB-17-08 Augmented Endoscopy System for the Detection of Mucosal Colorectal Polyps in Adult Patients Undergoing Screening or Surveillance Colonoscopy for CRC.
Brief Title: CB-17-08 Augmented Endoscopy System for Mucosal Lesion Detection During Colonoscopy for Colon Rectal Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmo Artificial Intelligence-AI Ltd (Industry)
Responsible Party: Sponsor
Organization: Cosmo Pharmaceuticals NV (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CB-17-08/03
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- With CB-17-08 CADe (Experimental)
  Interventions: Device: CB-17-08 CADe
- Without CB-17-08 CADe (No Intervention)

INTERVENTIONS:
Device: CB-17-08 CADe — CB-17-08 Augmented Endoscopy System with Computer Aided Detection (CADe) function
  Arms: With CB-17-08 CADe

SUMMARY:
The aim of this study is to assess the performance of the CB-17-08 to help endoscopists find potential mucosal polyps during the colonoscopy procedure, without significant noise disturbing the endoscopist attention, nor negative interference with the lesions detection than with the standard colonoscopy alone: the study will investigate whether the use of the device provides an increase in the number of adenomas per colonoscopy as compared to standard colonoscopy. The study will also evaluate the safety of the CB-17-08, assessing if the use of the system increases the total number of excisions without a commensurate number of adenomas as compared to standard colonoscopy.

DETAILED DESCRIPTION:
Study procedure:

Patients will be randomized (1:1) to one of the arms by an IWRS system. Randomization will be stratified by study endoscopist, to balance the number of patients randomized to either of the study groups (1:1) within the same endoscopist, by age (from to 45 to <65 years old; ≥65 years old) and by reason for colonoscopy (screening, surveillance <3 years from previous colonoscopy, surveillance 3-10 years from previous colonoscopy). Each endoscopist shall not enrol more than 90 patients.

The following study visits are foreseen for each patient:

Screening Visit A screening visit is performed at the investigational site. During this visit out-patients scheduled for colonoscopy will be informed about the aims, procedures, benefits and possible risks of the study prior to signing the informed consent form for inclusion in the study. Their medical history will be recorded as well as eventual clinical or laboratory examinations according to the local standard of care preparation for a colonoscopy, ) and the date for the colonoscopy procedure to be performed at the investigational site will be scheduled.

Tandem Colonoscopy Visit Each eligible patient returns to the clinic to undergo a same-day, back-to-back tandem colonoscopy examination performed by the same experienced endoscopist. The randomized allocation will determine whether patients will undergo standard high-definition white light colonoscopy with CB-17-08 immediately followed by standard high definition white light colonoscopy or standard high definition white light colonoscopy followed by standard high definition white light colonoscopy with CB-17-08.

Bowel preparation will be done according to the usual standard of care protocols of the individual sites. The quality of bowel preparation will be assessed during colonoscopy using the Boston Bowel Preparation Scale (BBPS). Sedation according to the sites best experience and standard procedures will be delivered to the patient by the endoscopist or an anaesthesiologist.

Subjects' vital signs (blood pressure [BP], hearth rate [HR] and oxygen saturation [SpO2]) will be measured and monitored prior to, during and at the end of the tandem colonoscopy procedure.

The endoscopist will be instructed to adhere to their usual withdrawal technique and to spend a minimum of 6 minutes withdrawing and examining the colonic mucosa. Time to reach the caecum and time to withdrawal from caecum to exit will be recorded for each colonoscopy. Clean withdrawal time, i.e. withdrawal time excluding the time spent for procedures or washings (if any), will be recorded. At least 6 minutes of clean withdrawal time will be required for all colonoscopies, in accordance to the current ASGE guideline. Withdrawal time, total procedure time, and time for pauses to allow polypectomies and biopsies to be performed will be recorded. Repeated examination of any of the colon segments (e.g. right colon) in normal modality or in retroflexion is not permitted.

Each colorectal polyp detected during the first procedure, as well as each polyp detected during the second procedure, will be immediately removed or biopsied and will be sent to the central histology laboratory for characterization. When a mucosal polyp is detected, its estimated size and morphological appearance according to Paris classification will be reported by the endoscopist on the CRF, as well as the anatomical location inside the colonic districts. On the basis of histological examination, polyps will be categorized according to revised Vienna classification and serrated lesion classification.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age: ≥45 years;
* Patients presenting to the endoscopy unit for a screening colonoscopy or a surveillance colonoscopy for CRC;
* Willingness to undergo tandem colonoscopies with and without the use of CB-17-08 on the same day and in the same procedural setting;
* Ability to provide written, informed consent and understand the responsibilities of trial participation;

Exclusion Criteria:

* The subject is pregnant or is planning a pregnancy during the study period;
* History of inflammatory bowel disease (IBD);
* History of colon resection;
* History of Familial adenomatous polyposis (FAP) syndrome or of Serrated Polyposis Syndrome (SPS);
* History of overt lower GI bleeding;
* History of colonic stricture;
* History of radiation therapy to the abdomen or pelvis;
* Patients with contraindications to colonoscopy such as presence of acute diverticulitis or toxic megacolon;
* Subjects with particular symptoms (e.g diarrhea) who, per clinical practice, have to undergo random biopsies in the colon.

Fecal Occult Blood Test (FOBT) or Fecal Immunochemical Test (FIT) positive patients will not be excluded from the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Adenoma miss rate [AMR] | Day 1
  AMR, defined as the number of histologically confirmed adenomas and carcinomas detected during the second colonoscopy divided by the total number of histologically confirmed adenomas and carcinomas detected during the first and second colonoscopy combined.

SECONDARY OUTCOMES:
Polyp Miss Rate [PMR] | Day 1
  PMR, defined as the number of histologically confirmed polyps detected during the second colonoscopy divided by the total number of histologically confirmed polyps detected during the first plus second colonoscopy combined.
  Diminutive (<5 mm) hyperplastic polyps of the rectosigmoid region will not be accounted for in the endpoint analysis.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Geisinger Medical Center, Danville, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Kansas City VA Medical Center, Kansas City, Kansas
  - Ascension St. John's Hospital, Detroit, Michigan
  - Mayo Clinic Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic La Crosse, La Crosse, Wisconsin
- ASL Roma 1 (Presidio Nuova regina Margherita), Roma, Italy
- United Kingdom (2):
  - Queen Alexandra Hospital, Cosham
  - Oxford University Hospitals, Oxford

REFERENCES:
- [Derived] Wallace MB, Sharma P, Bhandari P, East J, Antonelli G, Lorenzetti R, Vieth M, Speranza I, Spadaccini M, Desai M, Lukens FJ, Babameto G, Batista D, Singh D, Palmer W, Ramirez F, Palmer R, Lunsford T, Ruff K, Bird-Liebermann E, Ciofoaia V, Arndtz S, Cangemi D, Puddick K, Derfus G, Johal AS, Barawi M, Longo L, Moro L, Repici A, Hassan C. Impact of Artificial Intelligence on Miss Rate of Colorectal Neoplasia. Gastroenterology. 2022 Jul;163(1):295-304.e5. doi: 10.1053/j.gastro.2022.03.007. Epub 2022 Mar 15. PMID 35304117